CLINICAL TRIAL: NCT02137993
Title: A Multi-center, Randomized, Double Blind, Parallel, PhaseⅣ Trial to Evaluate the Efficacy and Safety of A-prexa Compared to Zyprexa in Patients With Schizophrenia, Schizophreniform Disorder and Schizoaffective Disorder
Brief Title: Efficacy and Safety of A-prexa Compared to Zyprexa in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_OLZ_401
Record Dates: First submitted 2014-05-11; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-prexa (Experimental): A-prexa 5, 10mg
  Interventions: Drug: Zyprexa
- Zyprexa (Active Comparator): Zyprexa 5, 10mg
  Interventions: Drug: A-prexa

INTERVENTIONS:
Drug: A-prexa — A-prexa 5-20 mg for 6 weeks
  Arms: Zyprexa
Drug: Zyprexa — Zyprexa 5-20 mg for 6 weeks
  Arms: A-prexa

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of A-prexa compared to Zyprexa in patients with schizophrenia, schizophreniform disorder and schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* 20 years to 65 years
* Schizophrenia patient with an acute exacerbation
* Understand the requirement of the study and voluntarily consent to participate in the study

Exclusion Criteria:

* Patients who have another psychiatric disorders
* Patients who have unstable medical conditions
* Patients who have clinically important abnormalities of liver function test (>2.5 fold of upper normal limit), ECG and vital sign at screening visit
* Uncontrolled diabetic patients (plasma glucose level is more than 126 mg/dl in fasting condition)
* Patients who have a history of an allergic reaction to olanzapine
* Patient who have no clinical response to take two or more different atypical anti-psychotics for more than 4 weeks.
* Patient who take clozapine within 12 weeks before screening visit

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 6 week in total PANSS score | 6 week

SECONDARY OUTCOMES:
Change from baseline at 1, 2, 4 and 6 week in total PANSS score. | 6 week
Responder to be decreased of 30% or more in PANSS total score from baseline at 6 week | 6 week
Change from baseline at 6 week in total CGI-S score | 6 week
Responder rate in CGI-I score of 'very much improved', 'much improved' and 'minimally improved' | 6 week